CLINICAL TRIAL: NCT06590142
Title: Investigating the Interaction of the Enteric Nervous System With the Extrinsic Nervous System and the Immune System in Children and Development of Cell Therapies for Hirschsprung's Disease
Brief Title: Hirschsprung's Advances; Working Towards Autologous tIssue therapIes
Acronym: HAWAII
Status: Recruiting | Type: Observational
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: 322649
Record Dates: First submitted 2024-02-22; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hirschsprung Disease
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Ganglionic samples, transition zone and aganglionic segments of bowel, addressing the following objectives: 1. Characterising neural progenitor cells in three HSCR bowel segments using transcriptomics analysis. 2. Analysing the composition of cultured neurospheres from three HSCR bowel segments using flow cytometry and qPCR. 3. Determining the differentiation potential of neural progenitor cells in neurosphere cultures by modulating key signalling pathways including Notch, Sonic Hedgehog and serotonin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hirschsprung's - Aganglionic: Bowel specimens will be taken from the aganglionic segment of bowel from children with Hirschsprung's disease
  Interventions: Procedure: Observational study of tissue specimens
- Hirschsprung's - Ganglionic: Bowel specimens will be taken from the ganglionic segment of bowel from children with Hirschsprung's disease
  Interventions: Procedure: Observational study of tissue specimens
- Control: Bowel specimens will be taken from the bowel from children who do not have Hirschsprung's disease who are undergoing bowel surgery
  Interventions: Procedure: Observational study of tissue specimens

INTERVENTIONS:
Procedure: Observational study of tissue specimens — No intervention will be made

SUMMARY:
Children with Hirschsprung's Disease (HSCR) have no normal nerve cells in the lower end of their bowel. This can cause babies to die if left untreated treated. Currently the part of bowel that doesn't have normal nerves is removed with an operation, but this can have long-term complications including needing a permanent bag on the tummy for poo (stoma). Because of this there is an urgent need for better treatments.

The investigators have found that children with HSCR have nerve stem cells throughout their bowel, even in the lower end where the nerves haven't grown normally. We can grow these stem cells in the laboratory to form balls of nerve cells (neurospheres). The investigators want to find out whether these neurospheres grow into the nerves that are needed for the bowel to work normally. First the investigators will see how the nerve stem cells from the lower end of the bowel grow compared to those from the normal bowel. Then the investigators will see if the neurospheres change when the investigators put them with medications that affect growth of bowel nerves.

At the end of this project the investigators hope to know whether the nerve stem cells at the lower part of the bowel in children with HSCR can turn into bowel nerve cells that might make the bowel work normally. The investigators also hope to know whether the investigators can use medications to make the stem cells turn into normal nerves, meaning that children with HSCR could avoid an operation and a stoma.

DETAILED DESCRIPTION:
The gastrointestinal (GI) tract is responsible for many functions essential to life such as digestion, absorption and excretion, all of which are under the control of its own intrinsic nervous system, the enteric nervous system (ENS). The ENS is part of the autonomic peripheral nervous system and provides the intrinsic innervation of the bowel - the submucosal and myenteric plexuses are the two networks that comprise the ENS and consist of bundles of enteric neurons and glia - the enteric ganglia that are connected by nerve fibres. The ENS is essential for the autonomic regulation of gastric motility and secretion.

Hirschsprung's disease (HSCR) is a gut motility disorder, affecting 1 in 5000 people worldwide. HSCR is characterised by the absence of ganglia and nerve fibres of the ENS to various extents of the bowel: 80% of cases affect the distal colon and internal anal sphincter, but 10% of cases have total colonic aganglionosis and 1% total intestinal aganglionosis. Between the ganglionic and aganglionic bowel there is a transition zone. The transition zone is abnormally innervated due to a reduced number of enteric ganglia.

Initial presentation of neonates with HSCR typically includes distal intestinal obstruction, with symptoms including abdominal distention or vomiting and/or failure to pass meconium within the first 48hrs of life. Children with HSCR can also have difficulty feeding, severe constipation, and symptoms of HSCR- associated enterocolitis (HAEC).

Due to its lack of ENS, the aganglionic region of HSCR bowel is tonically contracted. This results in constipation and without treatment is fatal. The current gold-standard treatment for HSCR is a surgical pull-through procedure in which the aganglionic region and TZ is resected in an attempt to restore normal function.

The investigators have previously demonstrated the presence of enteric nervous system progenitor cells (ENSPCs) in the aganglionic bowel of children with HSCR. ENSPCs have both a multipotent nature and proliferative capacity. There has been a significant amount of research into the feasibility of using ENSPCs to reduce or correct bowel dysmotility in mouse and rat models of ENS neuropathies. ENSPCs have commonly been cultured as neurospheres. Neurospheres are free-floating cultures of neural stem cells that also contain neurons and glia and in the case of enteric neurospheres, ENSPCs.

ENSPCs cultured in neurospheres have the potential to be used as an autologous therapy for HSCR which would avoid the risk of immune rejection and can be isolated from embryonic and postnatal mouse, rat and human tissue. Enteric neurospheres have been shown to contain cells expressing various progenitor, neuronal and glial markers. In our lab demonstrated that both embryonic mouse caecum derived neurospheres and postnatal human colonic neurospheres expressed, the proliferation marker BrdU and the neuronal subtype markers NOS and VIP showing that neurosphere cells were capable of proliferation and differentiation. This work was further explored in the investigators' group and neurospheres were cultured from tissue from the aganglionic bowel of patients with HSCR. This demonstration indicates the potential for autologous therapies using the patients' own aganglionic bowel due to the presence of progenitor cells that were capable of differentiation into different neuronal subtypes in vitro.

The transplantation of enteric neurospheres to aganglionic bowel has provided insight into the ability of such cells to rescue a model with a HSCR phenotype. Using ex vivo models of aganglionic tissue, multiple groups have demonstrated that transplanted neurospheres can integrate into tissue and differentiate into enteric glia and electrophysiologically active neurons.

Recently, the investigators have found that there is an interaction in the transition zone of children with HSCR between the intrinsic ENS and the extrinsic nerves of the aganglionic bowel. As the transition zone is also resected during surgery for HSCR, this could provide a source of ENSPCs to use for autologous transplantation. However, transition zone neurospheres have not yet been characterised. The investigators plan to include transition zone neurospheres in our investigation to determine whether these cells may be useful for transplantation. This forms part of our next set of experiments to investigate future therapies for HSCR.

The clinical outcomes of children with Hirschsprung's Disease have been poorly reported. Recently a core outcome set has been developed to help to standardise how children's outcomes are reported and to encourage reporting of patient's experiences as well as clinician's experiences. After pull-through 30% of patients suffering constipation or incontinence, with clear 'constipation' and 'rapid transit' phenotypes being evident. This may be caused by abnormal motility of the ganglionic region or by the fact that the aganglionic internal anal sphincter remains after surgery. Future therapies for HSCR aim to reduce long term morbidities associated with HSCR but a key part of this includes drawing together children's lived experience with the findings within the laboratory. The investigators are currently undertaking a study of the long-term outcomes of children and adults with Hirschsprung's Disease (REC: 18/NNW/0608) and this study offers an opportunity to combine clinician and patient reported data with immunohistochemical data.

ELIGIBILITY:
Inclusion Criteria:

• Any child undergoing therapeutic intestinal resection (but specifically those in which it is not necessary for all resected tissue to be sent for histopathological analysis, as no additional tissue will be removed for research purposes).

Exclusion Criteria:

• None

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any child undergoing therapeautic intestinal resection.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2034-03-01 (Estimated); Study Completion 2036-03-01 (Estimated)

PRIMARY OUTCOMES:
Successful optimisation of a scRNAseq protocol using dissociated human bowel cells | 01/03/2026
  SC RNA sequencing will be successfully carried out on every specimen in which it is undertaken

CONTACTS AND LOCATIONS:
Locations (1):
- Alder Hey Children's NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

DOCUMENTS (1):
  • Study Protocol (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT06590142/Prot_000.pdf